CLINICAL TRIAL: NCT00563355
Title: A Prospective Randomised Controlled Trial to Study the Effects of Recombinant Human Erythropoietin on the Progression of Atherosclerosis, Cardiovascular Function, Nutrition and Residual Renal Function in Pre-dialysis Chronic Renal Failure Patients
Brief Title: A Study to Evaluate Whether Correction of Anemia Using Recombinant Human Erythropoietin Reduces the Progression of Atherosclerosis and Cardiac Hypertrophy in Pre-dialysis Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The Hong Kong Society of Nephrology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE2000.241; HARECCTR0500004
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Disease; Kidney Diseases; Cardiovascular Diseases
Keywords: chronic kidney disease; cardiovascular disease
MeSH Terms: conditions — Chronic Disease; Kidney Diseases; Cardiovascular Diseases; Renal Insufficiency, Chronic | interventions — Erythropoietin

INTERVENTIONS:
Drug: erythropoietin

SUMMARY:
The primary aim of the study is to evaluate the effects of correction of anemia using erythropoietin on the progression of atherosclerosis and cardiac muscle thickening in patients with chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic renal failure with serum creatinine between 150umol/L and 800umol/L and at the same time Hb
* Patients with regression line of 1/serum creatinine versus time showing that they may not require dialysis within the coming 12 months
* Patients below the age of 75

Exclusion Criteria:

* Patients with valvular heart disease/congenital heart disease
* Patients with ischemic heart disease/history of myocardial infarction/coronary artery bypass surgery
* Patients with history of heart failure
* Patients with regression line of 1/serum creatinine versus time showing that the estimated date of end stage renal disease is within 12 months
* Patients with thalassemic trait or haemoglobinopathies
* Patients with underlying haematological malignancies
* Patients with active bleeding
* Patients with uncorrected iron or other vitamins deficiencies
* Patients with poor general condition

Max Age: 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2001-02; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
endothelial function and atherosclerosis | 6 month, 1 year
cardiac hypertrophy and cardiac function | 6 month, 1 year

SECONDARY OUTCOMES:
nutrition status | 6 month, 1 year
residual renal function | 6 month, 1 year
quality of life | 6 month, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Angela YM Wang, Dr, Principal Investigator — Department of Medicine & Therapeutics/Nephrology, Prince of Wales Hospital/ The Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280